CLINICAL TRIAL: NCT05339243
Title: Evaluating the Safety and Efficacy of the Probiotic Bifidobacterium Longum ES1 and the Post Biotic Heat-treated Bifidobacterium Longum ES1 (HT-ES1) on IBS Symptom Severity in Patients With Diarrhoea Predominant Irritable Bowel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vedic Lifesciences Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: ADM/211001/BLE/IBS
Record Dates: First submitted 2022-04-13; First posted 2022-04-21 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-09

CONDITIONS: Irritable Bowel Syndrome With Diarrhea

STUDY DESIGN:
Intervention Model Description: A randomised, double-blind, placebo-controlled, parallel-group multicentre study
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ES 1 (Active Comparator): Two capsules orally once daily after breakfast for 84 days
  Interventions: Other: ES 1
- HT ES1 (Active Comparator): Two capsules orally once daily after breakfast for 84 days
  Interventions: Other: HT ES1
- Placebo (Placebo Comparator): Two capsules orally once daily after breakfast for 84 days
  Interventions: Other: Placebo

INTERVENTIONS:
Other: ES 1 — Two capsules orally once daily after breakfast for 84 days
  Arms: ES 1
Other: HT ES1 — Two capsules orally once daily after breakfast for 84 days
  Arms: HT ES1
Other: Placebo — Two capsules orally once daily after breakfast for 84 days
  Arms: Placebo

SUMMARY:
Randomized controlled clinical study has been proposed to evaluate the safety and efficacy of ES1 probiotic strain and heat-treated ES1 postbiotic strain in individuals suffering from IBS-D.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged ≥18 to ≤ 65 years.
2. Participants diagnosed with diarrhoea-predominant irritable bowel syndrome (IBS-D) as per ROME IV criteria:

   i) Recurrent abdominal pain on average at least one day/week in the last three months, associated with two or more of the following criteria: Related to defecation Associated with a change in stool frequency (increase/decrease in frequency). Associated with a change in the form (appearance) of stool. ii) History of abnormal bowel movements predominantly diarrhoea (>25% of bowel movement categorised as stool form type 6 or 7 (diarrhoea) and <25% as stool form type 1 or 2 constipation) on BSFS).
3. Participants with an IBS-SSS score ≥ 175.
4. Participants who test negative for COVID-19 by Rapid Antigen Lateral Flow Test Device.
5. Participants who can comply and perform the procedures as per the protocol (consumption of study medications, biological sample collection procedures, and study visit schedule).

   Female participants who are willing to use acceptable contraceptives during the study duration.
6. Participants who are literate enough to understand the purpose of the study and their rights.
7. Participants who are able to give written informed consent and are willing to participate in the study.

Exclusion Criteria:

1. Participants diagnosed with anxiety as assessed by STAI-AD S- anxiety subscale score ≥ 40.
2. Gluten and/or lactose intolerant individuals.
3. Abnormal Thyroid Stimulating Hormone (TSH) value which is (< 0.4 to > 4.2 mIU/L).
4. Participants with uncontrolled type II diabetes mellitus defined as random blood glucose (RBG) > 199 mg/dL or fasting blood glucose (FBG) >125 mg/dL.
5. Participants with a body mass index (BMI) ≥ 30 kg/m2.
6. Presence of uncontrolled hypertension defined as systolic blood pressure (SBP) ≥ 140 mm Hg and/or diastolic blood pressure (DBP) ≥ 90 mm Hg.
7. Participants with a history of intake of antibiotics (Rifaximin, metronidazole, or any other), other probiotics, prebiotics, synbiotic, proton pump inhibitors, acid sequestrants (cholestyramine, Bile colestipol), FODMAP diet, and histamine H2- receptor antagonists/H2 blockers within six weeks prior to the screening day.
8. Participants with a history of daily intake of antidepressants (Tricyclic antidepressants, Selective serotonin reuptake inhibitors (SSRIs), and Selective serotonin-norepinephrine reuptake Inhibitors (SSNRIs)), clonidine, otilonium bromide, asimadoline, eluxadoline, diphenoxylate, antispasmodics including mebeverine and pinnaverium and anticholinergics within two weeks before the screening day.
9. Participants with a history of bariatric surgery or surgical resection of the stomach, small intestine, or large intestine.
10. Participants showing signs of bile acid malabsorption (BAM), as evident from the history of green colour or foul odour of the stool during the last month.
11. Participants with a history of or complications from malignant tumours.
12. Participation in other clinical trials in the last 90 days prior to screening
13. Active smokers or using any form of smokeless tobacco.
14. Participants with substance abuse problems (within two years) defined as:
15. Use of recreational drugs (such as cocaine, methamphetamine, marijuana, etc.)/Nicotine dependence.
16. High-risk drinking as defined by the consumption of four or more alcohol-containing beverages on any day or eight or more alcohol- containing beverages per week for women and five or more alcohol-containing beverages on any day or 15 or more alcohol- containing beverages per week for men.
17. Participants having clinically significant illnesses of cardiovascular, endocrine, immune, respiratory, hepato-biliary, kidney and urinary, haematological, musculoskeletal system and/or any inflammatory disorder, tumour, and other gastrointestinal diseases.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2022-04-21 (Actual); Primary Completion 2023-01-13 (Actual); Study Completion 2023-01-13 (Actual)

PRIMARY OUTCOMES:
Irritable Bowel Syndrome-Symptom Severity Scale | day 0, 28, 56, and 84
  To determine the efficacy of investigational products on the participants global assessment of gastrointestinal symptoms, as assessed by change in Irritable Bowel Syndrome-Symptom Severity Scale total score at the end of study from baseline compared to placebo.
  Each of these 5 items is scored on a visual analogue scale from 0 to 100. Therefore, the total score on the ranges from 0 to 500. Participants are asked to respond to each question on a 100-point visual analogue scale. The higher the scores, the more will be the severity of symptoms. Participants, if required, can be categorized as having mild (75-175), moderate (175-300),
  Higher the score is the worst outcome and lower the score is the betterment.

SECONDARY OUTCOMES:
Bristol Stool Form Scale | day 0, 28, 56, and 84
  At the end of days 28, 56, and 84, the percentage of participants transitioning to normal stool consistency (as demonstrated by weekly BSFS score reported as 3, 4, or 5) compared to baseline scores will be identified to evaluate the efficacy of IP in comparison to placebo.
Irritable Bowel Syndrome-Quality of Life | day 0, 28, 56, and 84
  Quality of life as assessed by change in Irritable Bowel Syndrome-Quality of Life.
  It is a 34-item questionnaire with each item rated on a 5-point scale (34-170), with increasing scores indicating the deteriorating quality of life (Appendix-III). However, to facilitate comparisons among various measures on a standardized scale, the summed scores will be transformed to a 0 - 100 scale ranging from 0 (poor quality of life) to 100 (maximum quality of life).
Abdominal Pain Severity-Numeric Rating Scale score. | day 0, 28, 56, and 84
  Abdominal pain severity as assessed by change in Abdominal Pain Severity-Numeric Rating Scale (APS-NRS) score.
  score ratings include 0 - None, 1 to 3 - Mild, 4 to 6 - Moderate, 7 to 9 - Severe, and 10
  = very severe.4
State-Trait Anxiety Inventory-Adults score. | day 0, 28, 56, and 84
  Mental health as assessed by change in State-Trait Anxiety Inventory-Adults (STAI-AD) score. The State-Trait Anxiety Inventory has 40 items, 20 allocated to each S-Anxiety and T-Anxiety sub-scales . The range of scores for each subtest is 20-80, the higher score indicating greater anxiety. A cut point of 39-40 has been suggested to detect clinically significant symptoms for the S-Anxiety scale
Vitals - blood pressure | day 0, 28, 56, and 84
  To evaluate the safety of IP consumption .
  Normal BP ranging Systolic120 - 129 mmHg and or diastolic 80 - 84 mm Hg
Gut microbiome as assessed by 16S rRNA sequencing of faecal samples. | day 0 and 84
Vitals - Pulse Rate | day 0, 28, 56, and 84
  Normal Pulse rate 60 - 100 bpm

CONTACTS AND LOCATIONS:
Locations (8):
- India (8):
  - Apex Gastro Clinic and Hospital, Ahmedabad, Gujarat
  - Gastroplus, Digestive disease centre, Ahmedabad, Gujarat
  - Aman Hospital and research centre, Vadodara, Gujarat
  - Shantaee Nursing Home, Mumbai, Maharashtra
  - Dr. Sanjeev Khanna clinic, Mumbai, Maharashtra
  - Stress test clinic, Mumbai, Maharashtra
  - Jaipur National University Institute for Medical Science & Research Centre, Jaipur, Rajasthan
  - Dr. Sudhir Maharshi clinic, Jaipur, Rajasthan

IPD SHARING:
Plan to Share IPD: Undecided